CLINICAL TRIAL: NCT01636947
Title: A Korean Multicenter, Randomized, Double-Blind, Clinical Trial to Evaluate the Efficacy and Tolerability of Aprepitant for the Prevention of Chemotherapy-Induced Nausea and Vomiting in the First Cycle of Moderately Emetogenic Chemotherapies (MEC, Non-AC Regimes) With Broad Range of Tumor Types (KMEC Study)
Brief Title: A Korean Study of Efficacy and Safety of Aprepitant-based Triple Regimen for the Prevention of Chemotherapy-Induced Nausea and Vomiting in the First Cycle of Moderately Emetogenic Chemotherapy (Non-doxorubicin Hydrochloride [Adriamycin] and Cyclophosphamide Regimens) (MK-0869-225) (KMEC)
Acronym: KMEC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0869-225; MK-0869-225 (Other: Merck protocol number)
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Results first posted 2015-07-30 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-08

CONDITIONS: Nausea; Vomiting
Keywords: chemotherapy; nausea; vomiting; emetogenic; cancer; antiemetics; tumor
MeSH Terms: conditions — Nausea; Vomiting; Neoplasms | interventions — Aprepitant; Ondansetron; Dexamethasone; dexamethasone 21-phosphate; dexamethasone acetate; Calcium Dobesilate; Granisetron; dolasetron; Tropisetron; Metoclopramide; alizapride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aprepitant Regimen (Experimental): Participants receive one aprepitant 125 mg capsule by mouth (PO) once daily (QD) on Day 1 and one aprepitant 80 mg capsule PO QD on Days 2 and 3 of Cycle 1. Participants also receive ondansetron 16 mg intravenously (IV) QD and dexamethasone 12 mg PO on Day 1 and placebo for ondansetron 8 mg PO twice daily (BID) on Days 2 and 3.
  Interventions: Drug: Aprepitant; Drug: Ondansetron; Drug: Dexamethasone; Drug: Ondansetron Placebo; Drug: Rescue Therapy (granisetron, dolasetron, tropisetron or ondansetron; metoclopramide or alizapride).
- Control Regimen (Active Comparator): Participants receive one placebo capsule PO QD on Day 1 and one placebo capsule PO QD on Days 2 and 3 of Cycle 1. Participants also receive ondansetron 16 mg IV QD and dexamethasone 20 mg PO on Day 1 and ondansetron 8 mg PO BID on Days 2 and 3.
  Interventions: Drug: Aprepitant Placebo; Drug: Ondansetron; Drug: Dexamethasone; Drug: Rescue Therapy (granisetron, dolasetron, tropisetron or ondansetron; metoclopramide or alizapride).

INTERVENTIONS:
Drug: Aprepitant — Aprepitant (125 mg PO, QD) on Day 1, Aprepitant (80 mg PO, QD) on Days 2 and 3
  Other Names: MK-0869; EMEND® PO
  Arms: Aprepitant Regimen
Drug: Aprepitant Placebo — Aprepitant Placebo (PO, QD) on Days 1, 2, and 3
  Arms: Control Regimen
Drug: Ondansetron — Ondansetron (16 mg, IV, QD) on Day 1 and/or ondansetron (8 mg PO BID) on Days 2 and 3
  Other Names: ZOFRAN®
Drug: Dexamethasone — Dexamethasone (20 mg or 12 mg, PO) on Day 1
  Other Names: dexamethasone sodium phosphate; dexamethasone acetate; Decadron; Dexasone; Diodex; Hexadrol; Maxidex
Drug: Ondansetron Placebo — Ondansetron Placebo (PO, BID) on Days 2 and 3
  Arms: Aprepitant Regimen
Drug: Rescue Therapy (granisetron, dolasetron, tropisetron or ondansetron; metoclopramide or alizapride). — Use of a rescue therapy for nausea and vomiting is permitted throughout the study. Permitted rescue therapies include a drug from among the following classes: 5-hydroxytryptamine (5-HT3) antagonists (granisetron, dolasetron, tropisetron or ondansetron), benzodiazepines, or benzamides (e.g., metoclopramide or alizapride).

SUMMARY:
This is an efficacy and safety study to compare aprepitant with ondansetron for the prevention of nausea and vomiting in the first cycle of moderately emetogenic chemotherapy (MEC) in participants with solid tumors. MECs include a number of commonly used cancer chemotherapeutic drugs including: oxaliplatin-based, irinotecan-based, and carboplatin-based regimens.

The primary hypothesis of this study is that the Aprepitant Regimen is superior to the Control (ondansetron) Regimen with respect to the percentage of participants with No Vomiting Overall (in the 120 hours following initiation of MEC) in participants with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed malignant disease
* Scheduled to receive a single dose of one or more of moderately emetogenic chemotherapeutic agents during Cycle 1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2 or Karnofsky score ≥60
* Predicted life span ≥4 months
* Laboratory values demonstrating adequate hematologic status
* Premenopausal females must not be pregnant or lactating and must agree to use effective birth control

Exclusion Criteria:

* Received chemotherapy within 6 months prior to starting on study drugs
* Scheduled to receive subsequent treatment due to a refractory response to first or second line chemotherapy
* Received an investigational drug within 30 days prior to starting on study drugs
* Radiation therapy to the abdomen or pelvis in the week prior to starting on study drugs
* Vomiting in the 24 hours prior to starting on study drugs
* Active infection (e.g., pneumonia) or any uncontrolled disease (e.g., diabetic ketoacidosis, gastrointestinal obstruction) except for malignancy
* Known hypersensitivity to Aprepitant (EMEND®), Dexamethasone or 5-HT3 receptor antagonists
* Presentation with gastrointestinal obstruction symptoms
* Symptomatic primary or metastatic central nervous system malignancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2012-12-12 (Actual); Primary Completion 2014-08-04 (Actual); Study Completion 2014-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Kim JE, Jang JS, Kim JW, Sung YL, Cho CH, Lee MA, Kim DJ, Ahn MJ, Lee KY, Sym SJ, Lim MC, Jung H, Cho EK, Min KW. Efficacy and safety of aprepitant for the prevention of chemotherapy-induced nausea and vomiting during the first cycle of moderately emetogenic chemotherapy in Korean patients with a broad range of tumor types. Support Care Cancer. 2017 Mar;25(3):801-809. doi: 10.1007/s00520-016-3463-0. Epub 2016 Nov 8. PMID 27826874
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0869-225&kw=0869-225&tab=access

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aprepitant Regimen | Control Regimen
Started | 244 | 250
Treated | 242 | 248
Completed | 232 | 239
Not Completed | 12 | 11
Not completed — Not Treated | 2 | 2
Not completed — Lost to Follow-up | 4 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Did Not Meet Eligibility Criteria | 1 | 4

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population consists of All Treated Participants. Two participants in each treatment group did not receive study drug.
Groups:
- Aprepitant Regimen: Participants receive one aprepitant 125 mg capsule PO QD on Day 1 and one aprepitant 80 mg capsule PO QD on Days 2 and 3 of Cycle 1. Participants also receive ondansetron 16 mg IV QD and dexamethasone 12 mg PO on Day 1 and placebo for ondansetron 8 mg PO BID on Days 2 and 3.
- Total: Total of all reporting groups
Arm/Group | Aprepitant Regimen | Control Regimen | Total
Number analyzed (Participants) | 242 | 248 | 490
Age, Customized [Number; unit: Participants]
  20 to 29 years | 4 | 3 | 7
  30 to 39 years | 5 | 10 | 15
  40 to 49 years | 32 | 28 | 60
  50 to 59 years | 73 | 65 | 138
  60 to 69 years | 74 | 77 | 151
  ≥70 years | 54 | 65 | 119
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 111 | 219
  Male | 134 | 137 | 271

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With No Vomiting - Overall Stage
Description: A vomiting episode was defined as one or more episodes of emesis (expulsion of stomach contents through the mouth) or retches (an attempt to vomit that is not productive of stomach contents). No vomiting during the Overall Stage was defined as no episodes of emesis during the 120 hours (Days 1-5) after initiation of moderately emetogenic chemotherapy (MEC).
Time Frame: Hour 0 on Day 1 to Day 5 (approximately 120 hours)
Population: The modified intention-to-treat (mITT) population consisted of all randomized participants who received chemotherapy, took ≥1 dose of study drug and had ≥1 post-treatment assessment on Day 1 and Day 2.
Measure: Number; unit: Percentage of Participants
Arm/Group | Aprepitant Regimen | Control Regimen
Number analyzed (Participants) | 237 | 243
Percentage of Participants | 77.2 | 72.0
Statistical Analysis 1: Comparison: Aprepitant Regimen vs Control Regimen; Test type: Superiority or Other; p = 0.191, Pearson's chi-square test

2. Secondary Outcome: Percentage of Participants With a Complete Response - Overall, Acute, and Delayed Stages
Description: A Complete Response was defined as no vomiting or dry heaves and no use of a rescue therapy. Overall Stage=0 to 120 hours after initiation of MEC. Acute Stage=0 to 24 hours after initiation of MEC. Delayed Stage=25 to 120 hours after initiation of MEC.
Time Frame: Hour 0 on Day 1 to Day 5 (approximately 120 hours)
Population: The mITT population consisted of all randomized participants who received chemotherapy, took ≥1 dose of study drug and had ≥1 post-treatment assessment on Day 1 and Day 2.
Measure: Number; unit: Percentage of Participants
Arm/Group | Aprepitant Regimen | Control Regimen
Number analyzed (Participants) | 237 | 243
Percentage of Participants
  Overall Stage | 73.4 | 70.4
  Acute Stage | 95.8 | 97.9
  Delayed Stage | 74.3 | 71.2
Statistical Analysis 1: Comparison: Aprepitant Regimen vs Control Regimen; Overall Stage p-value; Test type: Superiority or Other; p = 0.458, Pearson's chi-square test

3. Secondary Outcome: Number of Emetic Events - Overall Stage
Description: The number of emetic events that occurred during the Overall Stage (0 to 120 hours after initiation of MEC) are presented.
Time Frame: Hour 0 on Day 1 to Day 5 (approximately 120 hours)
Population: as for outcome 2
Measure: Number; unit: Number of Emetic Events
Arm/Group | Aprepitant Regimen | Control Regimen
Number analyzed (Participants) | 237 | 243
Number of Emetic Events | 54 | 68

4. Secondary Outcome: Percentage of Participants With No Vomiting and No Significant Nausea - Overall Stage
Description: Nausea was to be assessed using a 100-mm horizontal visual analogue scale (VAS) located in the participant diary labeled: "How much nausea have you had over the last 24 hours?" The left end of the scale (0 mm) was labeled "no nausea," and the right end of the scale (100 mm) is labeled "nausea as bad as it could be." In this study, No Significant Nausea was defined as a VAS nausea rating <25 mm.
Time Frame: Days 1 to Day 5
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Aprepitant Regimen | Control Regimen
Number analyzed (Participants) | 237 | 243
Percentage of Participants | 76.4 | 72.4

5. Secondary Outcome: Percentage of Participants With No Impact on Daily Life - Overall Stage
Description: The Functional Living Index-Emesis questionnaire (FLIE) is a validated, participant-reported instrument to measure the impact of chemotherapy-induced nausea and vomiting on daily life. There are 9 nausea-related items and 9 vomiting-related items, each on a 7-point scale. For the purposes of this study, "No Impact" on daily life was defined as an average item score of >6 on the 7-point scale; a total score >108 indicates no impact on daily life. Overall Stage=0 to 120 hours after initiation of MEC.
Time Frame: Day 6
Population: The mITT population consisted of all randomized participants who received chemotherapy, took ≥1 dose of study drug, had ≥1 post-treatment assessment on Day 1 and Day 2 and completed the FLIE questionnaire on Day 6.
Measure: Number; unit: Percentage of Participants
Arm/Group | Aprepitant Regimen | Control Regimen
Number analyzed (Participants) | 233 | 237
Percentage of Participants | 76.8 | 73.8

6. Secondary Outcome: Number of Participants With No Use of a Rescue Therapy - Overall, Acute, and Delayed Stages
Description: The percentage of participants who used no rescue therapy after initiation of MEC is presented for the Overall, Acute and Delayed Stages. Overall Stage=0 to 120 hours after initiation of MEC. Acute Stage=0 to 24 hours after initiation of MEC. Delayed Stage=25 to 120 hours after initiation of MEC.
Time Frame: Day 1 to Day 5
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Aprepitant Regimen | Control Regimen
Number analyzed (Participants) | 237 | 243
Percentage of Participants
  Overall Stage | 84.8 | 87.7
  Acute Stage | 98.7 | 99.2
  Delayed Stage | 84.8 | 88.5

7. Secondary Outcome: Percentage of Participants With One or More Clinical Adverse Event
Description: An adverse event was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the study drug. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition, which is temporally associated with the use of the study drug, is also an adverse event. Nausea and vomiting experienced during Days 1-6 were not counted as adverse events unless they were reported as a serious adverse event.
Time Frame: Day 1 through Day 29 (Up to 28 days after first dose of study drug)
Population: All randomized participants who received chemotherapy and took ≥1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Aprepitant Regimen | Control Regimen
Number analyzed (Participants) | 242 | 248
Percentage of Participants | 56.2 | 53.2

8. Secondary Outcome: Percentage of Participants With No Vomiting - Acute and Delayed Stages
Description: A vomiting episode was defined as one or more episodes of emesis (expulsion of stomach contents through the mouth) or retches (an attempt to vomit that is not productive of stomach contents). Acute Stage=0 to 24 hours after initiation of MEC. Delayed Stage=25 to 120 hours after initiation of MEC.
Time Frame: Day 1, Day 2 to Day 5
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Aprepitant Regimen | Control Regimen
Number analyzed (Participants) | 237 | 243
Percentage of Participants
  Acute Stage | 95.8 | 98.8
  Delayed Stage | 78.5 | 72.4

ADVERSE EVENTS:
Time Frame: Up to 28 days after first dose of study drug (Up to 29 days)
Description: The safety population consisted of all randomized participants who received chemotherapy and took ≥1 dose of study drug. Nausea and vomiting experienced during Days 1-6 were not counted as adverse events unless they were reported as a serious adverse event.
Arm/Group | Aprepitant Regimen | Control Regimen
Serious Adverse Events (participants affected / at risk) | 25/242 | 16/248
Other Adverse Events (participants affected / at risk) | 87/242 | 96/248
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aprepitant Regimen (N=242) | Control Regimen (N=248)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Menopausal symptoms (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Neutropenic colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (1)
Asthenia (General disorders) | 3 (3) | 1 (1)
Catheter site pain (General disorders) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (4) | 3 (3)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Wound dihiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aprepitant Regimen (N=242) | Control Regimen (N=248)
Constipation (Gastrointestinal disorders) | 10 (10) | 22 (22)
Diarrhoea (Gastrointestinal disorders) | 14 (15) | 17 (17)
Nausea (Gastrointestinal disorders) | 20 (20) | 20 (20)
Neutrophil count decreased (Investigations) | 22 (22) | 21 (21)
Decreased appetite (Metabolism and nutrition disorders) | 14 (15) | 15 (15)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (11) | 18 (18)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 6 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (9) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this study 60 days prior to submission for publication/presentation.